CLINICAL TRIAL: NCT04300699
Title: Feasibility of Frailty Assessment and Implementation of Protocol-led Geriatric Interventions in Women Over the Age of 70 With Epithelial Ovarian Cancer in the Oncology Clinic (FAIR-O)
Brief Title: Feasibility of Frailty Assessment and Implementation of Interventions in Women Over 70 With Epithelial Ovarian Cancer
Acronym: FAIR-O
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CCR 5138; RG2165 (Other Grant/Funding Number: Wellbeing of Women)
Record Dates: First submitted 2020-03-02; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2019-11

CONDITIONS: Ovarian Cancer; Chemotherapy; Quality of Life; Tolerance; Aged
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Single cohort intervention design with 12 month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovarian cancer patients over 70 years receiving chemotherapy (Other): Patients with ovarian cancer receiving chemotherapy as either first line treatment (i.e. newly diagnosed advanced stage III/IV cancer) or at first relapse. Patients to receive a Geriatric Assessment including interventions for functional or other identified deficits and appropriate specialist algorithm-determined interventions.
  Interventions: Other: Functional Geriatric Assessment

INTERVENTIONS:
Other: Functional Geriatric Assessment — A series of 8 self-completed questionnaires for the identification of functional deficits which will be addressed via algorithm-guided interventions and assessments.

SUMMARY:
Ovarian cancer is frequently diagnosed in older women, with over half of all new diagnoses being in women over 65 years. Current treatment options are based on the results of clinical trials that often do not include older, less fit patients in whom treatments may be less well tolerated. Further, in older patients the impact of complex medical and social issues is not known. The UK lags behind Europe and the United States in the development of research programs dedicated to improving outcomes for older patients. More research focus is urgently required to improve the assessment and management of older women with ovarian cancer to improve survival outcomes, quality of life and functional independence.

Current treatment decisions are made predominantly on age and fitness. However, it has been shown that undertaking a holistic, geriatric assessment of older patients can highlight important issues that would not necessarily be identified in a routine oncology appointment. In this study, we propose to ask oncology teams to undertake a geriatric assessment and specifically address issues that may arise as a result of this. The assessment comprises 8 simple non-invasive assessments that can be performed in the out-patient setting.

This approach could result in an important change in clinical practice leading to more holistic assessment of older cancer patients and better address their specific needs and manage their cancer treatment. The long-term goal is to show that pro-actively managing potential issues at the beginning of treatment allows patients to tolerate treatment and maintain their functional independence, leading to improved quality of life.

DETAILED DESCRIPTION:
FAIR-O is a single-arm, multi-center, phase II intervention trial of a geriatric assessment in older patients (≥ 70 years old) diagnosed with epithelial ovarian, fallopian tube or primary peritoneal cancer. Patients will be approached if they are being considered for systemic chemotherapy either as neoadjuvant / front-line chemotherapy in the first-line setting OR for chemotherapy at first relapse.

Two cohorts of patients will be recruited and run in parallel (no comparison will be performed between them):

1. First-line cohort: patients with newly diagnosed advanced (stage III/IV) ovarian cancer who have received no prior treatment for ovarian cancer including surgery.
2. First relapse cohort: ovarian cancer patients with first relapse

On consenting to the trial, a comprehensive medical and treatment history will be obtained including blood tests, tumour markers and a CT scan. The CT scan will be assessed for extent (volume) of muscle mass and compared to reference standards to identify patients with low muscle attenuation and sarcopenia (i.e. loss of muscle mass).

In addition, consented patients will be asked to undertake a comprehensive Geriatric Assessment which comprises a collection of 8 tests - all of which are non-invasive. These test comprise validated questionnaires and functional assessments including the G8 questionnaire, independent activities of daily living (IADL), activities of daily living (ADL), Charlson co-morbidity score, Hospital anxiety and depression scale (HADS), mini nutritional assessment (MNA), a timed up-and-go test and a mini cognitive assessment.

The Geriatric Assessment will enable the treating clinical team to determine whether the patient has specific deficits or problems which need further specialist attention with the aim of ensuring maximum tolerance to chemotherapy treatment. A Study Algorithm will guide the clinician to the most appropriate actions. These actions may include referral to other specialist services or referral for specific diagnostic tests. The number and type of referrals and the time taken for that referral to be performed will be captured.

Following the initial assessment in clinic, patients will will continue to attend standard treatment chemotherapy clinics. Their response to treatment will be recorded including the emergence of symptoms of study interest. Throughout the study decisions regarding systemic chemotherapy including regimen choice, dose modifications and supportive medications will be the responsibility of the treating oncologist and will not be determined by the outcome of the Geriatric Assessment.

Patients will be recruited until 60 patients have been recruited to each cohort. Patients will be followed-up until the end of the study which will be defined as 12 months from study entry or disease progression or death, whichever comes soonest.

The feasibility of introducing the Geriatric Assessment into the standard of care chemotherapy pathway is the primary end point of the study and will be statistically assessed. The number of fully completed assessments that the Research Team are able to conduct in the predicted target of 120 patients recruited to the trial will determine the feasibility on introducing the Geriatric Assessment to routine oncology clinics for this patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age at time of consideration for systemic chemotherapy of 70 years and above
* Histological or cytological confirmation of epithelial ovarian cancer
* Planning to commence systemic chemotherapy for either newly diagnosed epithelial ovarian cancer or first disease relapse
* Life expectancy greater than 3 months
* Able to give informed consent, complete questionnaires in english and comply with study procedures

Exclusion Criteria:

* In the opinion of the investigator, patient is not fit for systemic chemotherapy or patient declines systemic chemotherapy
* Patient does not have the capacity to consent for enrollment into the study or capacity to consent for systemic chemotherapy

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of completing the Functional Geriatric Assessment | Obtained at Baseline (Date of Consent)
  Proportion of patients in whom it was possible to complete the Functional Geriatric assessment within the Oncology Clinic setting, assessed at the point of the first oncology clinic visit.

SECONDARY OUTCOMES:
Proportion of patients with deficits identified resulting in algorithm defined interventions | Obtained at Baseline (Date of Consent)
  The number of deficits identified through use of the Functional Geriatric Assessment resulting in algorithm defined interventions including clinical referrals or assessments as identified during the first oncology clinic visit.
Proportion of patients developing sarcopenia during chemotherapy treatment, amounting to an average of 6 months on chemotherapy treatment. | Baseline (Date of Consent) to date of last chemotherapy treatment, an average of 6 months.
  The number of patients assessed as sarcopenic as assessed via routine computerized tomography scans conducted at baseline, mid-treatment and the end of treatment.
Proportion of patients with grade 3/4 hematological and non-hematological toxicities | Baseline (date of Consent) to date of last chemotherapy treatment, an average of 6 months.
  The number of patients experiencing Grade 3 or 4 hematological and non-hematological toxicities using the Common Terminology Criteria for Adverse Events (CTCAE) assessed through chemotherapy treatment from the start of treatment, mid-way through treatment and at the end of treatment, an average time-frame of 6 months.
Time on chemotherapy treatment | Start date of chemotherapy treatment to date of discontinuation of treatment, an average of 6 months.
  The length of time in months and days that the patient remains on routine chemotherapy treatment, an average of 6 months.
Quality of Life Outcome score in Cancer Patients | Start date of chemotherapy treatment, through treatment (average of 6 months) and at months 3, 6, 9, and 12 after date of last delivery of chemotherapy treatment.
  Quality of Life measured using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30. Maximum (worst) score: 112 and minimum (best) score: 28
Quality of Life Outcome score in Ovarian Cancer Patients | Start date of chemotherapy treatment, through treatment (average of 6 months) and at months 3, 6, 9, and 12 after date of last delivery of chemotherapy treatment.
  Quality of Life measured using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire in Ovarian Cancer Patients (QLQ OV) 28. Maximum (worst) score: 112 and minimum (best) score: 28
Quality of Life Outcome score in Elderly Cancer Patients | Start date of chemotherapy treatment, through treatment (average of 6 months) and at months 3, 6, 9, and 12 after date of last delivery of chemotherapy treatment.
  Quality of Life measured using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire in Elderly Cancer Patients (QLQ ELD) 14. Maximum (worst) score: 56 and minimum (best) score: 14
Sarcopenia and frailty | Assessed between baseline (date of Consent) mid-way though chemotherapy treatment to the date of delivery of last chemotherapy treatment, an average of 6 months.
  Sensitivity and specificity of sarcopenia in identifying frailty as identified by the Functional Geriatric Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Susana Banerjee, MBBS MA FRCP, Principal Investigator — Royal Marsden NHS Foundation Trust